CLINICAL TRIAL: NCT05036031
Title: Liver Transplantation for EASL-CLIF and APASL ACLF Patients: a Retrospective Cohort Study to Evaluate Different Criterion in Predicting Post-transplant Outcomes
Brief Title: Transplantation for EASL-CLIF and APASL ACLF Patients: a Retrospective Cohort Study
Acronym: TEA-ACLF
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Renji-IIT2021091
Record Dates: First submitted 2021-09-01; First posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Acute-On-Chronic Liver Failure; Liver Cirrhosis; Liver Transplant; Complications
Keywords: Acute-On-Chronic Liver Failure; EASL-CLIF criteria; APASL criteria
MeSH Terms: conditions — Acute-On-Chronic Liver Failure; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- EASL-CLIF ACLF patients
- APASL ACLF patients
- Non-ACLF patients

SUMMARY:
The definition and diagnostic criteria of acute-on chronic liver failure (ACLF) differed evidently between the East and the West due to the difference in the underlying etiology. Liver transplantation is the most effective treatment to reverse the progress of ACLF and improve the survival rate of patients. The purpose of this study is to explore the accuracy of the two diagnostic criteria of EASL-CLIF and APASL ACLF in assessing the survival rate of patients with liver cirrhosis after LT.

DETAILED DESCRIPTION:
A retrospective collection and analysis of the preoperative conditions of patients with LT due to cirrhosis in a single center from January 2015 to June 2020 would be conducted, including epidemiological characteristics, etiology, clinical indicators, and short-term (28 days, 90 days) and long-term (1 year, 3 years) survival after LT.

ELIGIBILITY:
Inclusion Criteria:

* patients underwent liver transplantation for cirrhosis
* The diagnosis of ACLF followed APASL and EASL-CLIF definition.

Exclusion Criteria:

* Patients with malignant tumor or underwent living donor liver transplantation (LDLT) were excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients underwent liver transplantation for cirrhosis at Renji Hospital, School of Medicine, Shanghai Jiao Tong University, China between January 2015 and June 2020 were considered for inclusion.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
3 years overall survival | Up to ~3 years

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Xia, Study Chair — Dept. Liver Surgery, Renji Hospital, School of Medicine, SJTU; Hao Feng, Principal Investigator — Ren Ji Hospital, School of Medicine, Shanghai Jiao Tong University